CLINICAL TRIAL: NCT04896489
Title: Neuroimaging Mechanisms by Which Memory and Glucocorticoids Promote Risky Drinking
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2000026404
Record Dates: First submitted 2021-05-17; First posted 2021-05-21 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-06

CONDITIONS: Alcohol Drinking; Drinking Behavior; Episodic Memory; Long-term Memory
MeSH Terms: conditions — Alcohol Drinking; Drinking Behavior | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- hydrocortisone (Experimental): Participants receive hydrocortisone (20mg)
  Interventions: Drug: Hydrocortisone 20 MG
- placebo (Placebo Comparator): Participants receive placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Hydrocortisone 20 MG — Participants receive Hydrocortisone 20 MG
  Arms: hydrocortisone
Other: Placebo — Participants receive placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to determine whether hydrocortisone biases formation of alcohol-related memories to potentiate drinking.

DETAILED DESCRIPTION:
This study aims to 1) Characterize the effect of elevated glucocorticoids during encoding on long-term memory for alcohol-related information; 2) Identify the neural mechanisms by which glucocorticoids influence encoding of alcohol-related experiences; and 3) Determine how glucocorticoid modulation of alcohol-related encoding relates to drinking after retrieving alcohol-related memories.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and write English
* BMI 18-35
* Beer drinking

Exclusion Criteria:

* Meet current criteria for any substance use disorder, excluding caffeine
* Current significant medical conditions or psychiatric symptoms requiring medication
* Current use of medications/drugs that interfere with the HPA axis response
* Peri and post-menopausal women, pregnant or lactating women, and those with hysterectomies
* Metal in body (for MRI safety)
* Systemic fungal infections (contraindication for hydrocortisone)
* Known hypersensitivity to components of hydrocortisone tablets (hydrocortisone, calcium stearate, corn starch, lactose, mineral oil, sorbic acid, sucrose)

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Changes fMRI signal | 1 hour
  Changes in fMRI signal at encoding will be assessed over an hour long period.
Item memory | Up to 90 minutes
  Item memory will be assessed through performance on delayed memory assessments. Item memory is determined by the accuracy of memory for individual items and will be expressed as dprime.
Context memory | Up to 90 minutes
  Context memory will be assessed through performance on delayed memory assessments. Context memory is determined by the accuracy of memory for associated contexts and will be expressed as % correct.
Affect memory | Up to 90 minutes
  Affect memory will be assessed through performance on delayed memory assessments. Affect memory is determined by subjective ratings of vividness (1-4), change in ratings from encoding to retrieval of memory (0-3). The score is averaged where a higher score indicates greater affect.

SECONDARY OUTCOMES:
Alcohol motivation | 10 minutes
  Performance on alcohol taste test following memory retrieval will be assessed using the Alcohol Taste Test (ATT). The test asks participants to taste the alcohol in each two containers to identify whether the alcohol was the same or different. The % correct is used to assess this outcome.
Affect - Negative | 10 minutes
  Self-reported measures of emotional state following drug administration and memory retrieval using the PANAS. The negative subscale of the PANAS will be used and has a range of 10-50. Higher scores indicate higher negative affect.
Affect - Positive | 10 minutes
  Self-reported measures of emotional state following drug administration and memory retrieval using the PANAS. The negative subscale of the PANAS will be used and has a range of 10-50. Higher scores indicate higher positive affect.
Neuroendocrine/cortisol reactivity | Baseline to 2 hours
  Change in salivary cortisol levels following the hydrocortisone/placebo administration.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth V Goldfarb, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in published articles will be shared after de-identification.
Supporting Information: Study Protocol
Time Frame: Immediately following publication with no end date.
Access Criteria: Anyone who wishes to have access to the data may do so.